CLINICAL TRIAL: NCT06048393
Title: A Phase I Clinical Study of Novel Coronavirus Broad-spectrum Neutralizing Antibody SA55 Nasal Spray in Healthy People
Brief Title: SA55 Novel Coronavirus Broad-spectrum Neutralizing Antibody Nasal Spray in Health People
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-SA55-1002
Record Dates: First submitted 2023-08-26; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): Single-dose:1 spray per side per time, 1ml/time Single-dose: 2 sprays per side per time, 2ml/time Multi-dose:1 spray per side per time, 1ml/time Multi-dose: 2 sprays per side per time, 2ml/time
  Interventions: Drug: SA55 nasal spray
- Group2 (Placebo Comparator): Single-dose: 1 spray per side per time Multi-dose: 2 sprays per side per time
  Interventions: Drug: SA55 nasal spray

INTERVENTIONS:
Drug: SA55 nasal spray — The novel coronavirus broad-spectrum neutralizing antibody SA55 nasal spray (SA55 nasal spray) is provided by Beijing Kexing Zhongwei Biotechnology Co., Ltd. The main component of this product is the novel coronavirus broad-spectrum neutralizing antibody, which is a colorless to pale yellow solution. Each milliliter contains 5mg of broad-spectrum neutralizing antibody against novel coronavirus. Excipients include histidine hydrochloride, arginine hydrochloride, histidine, sucrose, polysorbate 80 (II), hydroxypropyl cellulose, glycerol, and benzalkonium chloride (concentration 0.005%).
  20 sprays per bottle, approximately 100 sprays per bottle μ L. Containing 0.5 mg of broad-spectrum neutralizing antibody against novel coronavirus.

SUMMARY:
To evaluate the safety, tolerance, local drug content and neutralization activity in nasal cavity, systemic exposure level and immunogenicity of novel coronavirus broad-spectrum neutralizing antibody SA55 nasal spray.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65 on the day of enrollment;
* Overall good health condition, with no significant abnormalities during screening and/or pre medication physical examinations;
* Male subjects weighing ≥ 50.0kg; Female subjects with a weight of ≥ 45.0kg and a BMI between 18.0-28.0kg/m2 (including boundary values);
* The subjects (males and females with fertility potential) and their sexual partners have no fertility plan from 4 weeks before screening to 3 months after the last administration of the investigational drug, voluntarily take effective contraceptive measures, and have no plans to donate sperm or eggs;
* Volunteer to participate in the experiment, cooperate with the visit, and sign an informed consent form before the start of the study.

Exclusion Criteria:

* Individuals who are known to be allergic to the investigational drug, any component in the preparation, or other similar drugs;
* Individuals with a history of severe allergies or sensitivity to inhaled allergens, including but not limited to allergic rhinitis, bronchial asthma, etc;
* Previous history of sinus and septum surgery or radiotherapy;
* Patients with nasal diseases that may affect the deposition/absorption of drugs in the nose (such as narrowing of the nasal vestibule, severe deviation, perforation, ulcer of the nasal septum, thickening, pallor, edema, erosion of the nasal mucosa, hypertrophy and atrophy of the nasal wings, accumulation of fluid and pus in the nasal cavity, and space occupying or vegetation in the nasal cavity);
* Abnormal examination of the oropharynx has clinical significance, such as congestion, thickening, ulcers, hyperplasia or nodules, new organisms or foreign bodies of the throat mucosa;
* The following symptoms or diseases with clinical significance: a) a history of long-term nasal congestion, runny nose, headache, nosebleed, and other symptoms; b) Asthma, chronic respiratory diseases, etc; c) History of allergic rhinitis, chronic rhinitis, and sinusitis; d) History or signs of nasal, pharyngeal, and upper respiratory diseases that other researchers believe may affect the interpretation of the research process and/or local adverse events;
* Suffering from severe neurological disorders (epilepsy, seizures or convulsions) or mental illness, with a family history of mental illness, and neurological and psychiatric problems associated with various organic disorders;
* Abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities) or obvious bruising or coagulation disorders diagnosed by a doctor;
* Other uncontrolled chronic or severe disease history, including but not limited to cardiovascular disease, hematological system disease, liver and kidney disease, digestive system disease, respiratory system disease, malignant tumor, history of major organ transplantation, HIV/HBV/HCV/syphilis infection, or any other disease or physiological condition that the researcher believes can interfere with the test results;
* Planned pregnancy within 3 months, already pregnant (including positive pregnancy test), or breastfeeding;
* Received any SARS-CoV-2 neutralizing antibody injection that has been marketed or under research within 180 days prior to screening, or participated in clinical trials of other drugs or medical devices within 90 days prior to screening;
* Individuals who are unable to cooperate with nasal spray inhalation, nasal swab sampling, and venous blood collection, or who require long-term/intermittent use of any nasal products;
* Those with a body temperature above 37.0 ℃ before the first medication;
* 4 weeks prior to screening for clinically significant acute or chronic disease exacerbations, or a history of surgery;
* Known to have a history of SARS-CoV-2 infection within 3 months;
* Within 90 days before the first medication, blood donation>400 mL or significant blood loss>400 mL; Or donate plasma within 30 days before the first medication;
* Within 180 days prior to screening, use of immunoglobulins or blood products, immune modulators (such as adrenocortical hormones and thymosin) α Or blood stimulating drugs;
* Have been inoculated with any marketed or under research COVID-19 nasal spray vaccine within 180 days before screening, or have been inoculated with any marketed or under research COVID-19 vaccine within 90 days;
* Received attenuated live vaccine within 14 days prior to screening, or received subunit or inactivated vaccine within 7 days;
* Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, and functional vitamins within the first 14 days of screening;
* Smokers who smoke ≥ 5 cigarettes per day within the first 3 months of screening, or who cannot guarantee giving up smoking during the trial period;
* Drinking more than 14 units (1 unit of alcohol is equivalent to 360 mL of beer, 150 mL of wine, or 45 mL of Baijiu) per week within 3 months before screening, or not abstaining from alcohol during the test, or having a history of alcohol abuse within 2 years, or positive alcohol breath test before enrollment;
* There is a history of drug abuse or dependence or recreational drug use within 2 years prior to screening, or a positive urine drug abuse screening before enrollment.
* According to the judgment of the researchers, the subjects have any other factors that are not suitable for participating in clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SA55 nasal spray | 1 month
  The incidence and types of adverse events during the study period

SECONDARY OUTCOMES:
To evaluate the local drug content and neutralization activity in the nasal cavity at different time points after single and multiple administration of SA55 nasal spray | 1 month
  The local drug content in the nasal cavity at different time points after single and multiple administration
To evaluate the systemic exposure level of SA55 nasal spray after single and multiple administration | 1 month
  Concentration of SA55 in serum at different time points after medication

CONTACTS AND LOCATIONS:
Overall Officials: Ronghua Jin, M.D., Principal Investigator — Beijing Ditan Hospital
Locations (1):
- Beijing Ditan Hospital Capital Medical University, Beijing, Chaoyang, China

IPD SHARING:
Plan to Share IPD: Undecided